CLINICAL TRIAL: NCT02258932
Title: Eating Behaviours, Quality of Life and Cardiometabolic Risks in Adults With Type 1 Diabetes Using Continuous Subcutaneous Insulin Infusion Therapy - A Longitudinal Study
Brief Title: CSII in Type 1 Diabetes: Diet, Quality of Life & Cardiometabolic Risks - A Longitudinal Study
Status: Completed | Type: Observational
Sponsor: Liverpool John Moores University (Other)
Collaborators: Liverpool University Hospitals NHS Foundation Trust (Other Government)
Responsible Party: Principal Investigator, Mr Richard Webb, Postgraduate Research Student, Liverpool John Moores University
Other Study IDs: 13/NW/0122-1
Record Dates: First submitted 2014-10-03; First posted 2014-10-08 (Estimated); Last update posted 2016-02-19 (Estimated); Status verified 2015-07

CONDITIONS: Type 1 Diabetes
Keywords: Type 1 diabetes; CSII; Continuous subcutaneous insulin infusion; Insulin pump; Nutrition; Eating behaviours; Quality of life; Cardiometabolic risks; Liverpool; NHS; Metabolomics; Observational; Lipoproteins; Lipids; Food; Food diary; Longitudinal
MeSH Terms: conditions — Diabetes Mellitus, Type 1

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 12 Months
Biospecimen Retention: Samples Without DNA — Plasma will be retained for use by the research team during the study. After the study remaining samples will be destroyed in accordance with the Human Tissue Authority Code of Practice.
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Continuous subcutaneous insulin infusion: This group will consist of patients with Type 1 diabetes commencing continuous subcutaneous insulin infusion therapy.

SUMMARY:
Glycaemic control is an important aspect of Type 1 diabetes (T1D) management for diabetologists and patients alike. Evidence suggests continuous subcutaneous insulin infusion (CSII) is an effective method of achieving this. Among the advantages of CSII is the opportunity for patients to potentially discard relatively inflexible mealtimes and carbohydrate requirements imposed by other regimes such as multiple daily injections (MDI). There are also reported improvements in quality of life. Furthermore, in patients with good glycaemic control, such as those often assisted by CSII, various qualitative atherogenic lipid abnormalities may exist, despite the presence of a normal quantitative lipid profile; potentially leading to increased cardiometabolic risks. Literature examining the eating behaviours, quality of life and cardiometabolic risks of CSII patients over time after commencement of the therapy is sparse, frequently dated and worthy of further research.

DETAILED DESCRIPTION:
Continuous subcutaneous insulin infusion (CSII) is a therapy for patients with Type-1 diabetes mellitus involving insulin administration via electronic pump. CSII has been shown to reduce HbA1c levels and improve blood sugar control and the continuous, unobtrusive insulin delivery may potentially allow patients increased dietary flexibility and quality of life. However, despite these claims longitudinal investigatory literature is sparse. This study will clarify whether adult CSII patients experience eating behaviour and quality of life alterations over time after commencement of the therapy. This is important as changes may be associated with cardiometabolic risk variations; which will also be investigated.

Participants will comprise of a convenience sample of adults with Type-1 diabetes invited from diabetes clinics at the Royal Liverpool University Hospital who are due to commence CSII.

Following ethical consent the participants who are due to commence CSII will be observed at 5 time points (every three months) over a year. It should be noted that the recruitment period for the longitudinal arm of the study will be 9 months starting from the date the first participant is recruited. At each time point each participant will be asked to complete a 5 day food diary, a food intake questionnaire (FIQ), a quality of life (QOL) questionnaire, a semi-structured interview and give a 20ml sample of blood. This will be taken at the same time and in addition to their regular diagnostic sample, however where this is unfeasible extra occasional appointments may be needed. Results will be compared with existing patient medical records, which will also be analysed during the study.

ELIGIBILITY:
Inclusion Criteria:

* Patients must reside in Liverpool or the surrounding areas.
* Patients must be ages over 18
* Patients must have Type 1 diabetes
* Patients must be using or pending the supply of an insulin pump.

Exclusion Criteria:

* Patients must not live outside of Liverpool and the surrounding areas.
* Patients must not be aged under 18

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients will be selected from the Diabetes Centre from the Royal Liverpool and Broadgreen Hospital.
Sampling Method: Non-Probability Sample
Enrollment: 5 (Actual)
Dates: Start 2013-12; Primary Completion 2015-10 (Actual); Study Completion 2015-10 (Actual)

PRIMARY OUTCOMES:
Eating behaviours of adult patients with Type 1 diabetes using continuous subcutaneous insulin infusion therapy measured using food diaries and food surveys. | 12 months after commencement of the therapy.
  The primary outcome will be measured for 12 months using a combination of food intake questionnaires and food diaries.

SECONDARY OUTCOMES:
Quality of life of adults with Type 1 diabetes who are using insulin pump therapy. | 12 months after commencement of the therapy
  Quality of life will be assessed using a combination of semi-structured interviews and quality of life questionnaires.
Cardiometabolic risks of adult patients with Type 1 diabetes who are using insulin pump therapy. | 12 months after commencement of the therapy
  Cardiometabolic risks will be measured by accessing patient's medical records and taking a sample blood which will be analysed for lipoprotein subfractions, apolipoproteins (A1, A2 and B), HDL, LDL, NEFA, triglycerides and total cholesterol. Metabolomics analysis will also be carried out on collected plasma samples with a focus on both previously identified markers of cardiovascular disease and novel biomarkers.

CONTACTS AND LOCATIONS:
Overall Officials: Richard J Webb, BA, Principal Investigator — Liverpool John Moores University
Locations (1):
- Royal Liverpool and Broadgreen University Hospital, Liverpool, Merseyside, United Kingdom